CLINICAL TRIAL: NCT01560663
Title: Predictors of Response to Neoadjuvant Docetaxel-Carboplatin Chemotherapy for Patients With Stage II and III Triple Negative Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Miguel Martín Jiménez (Other)
Collaborators: UNC Lineberger Comprehensive Cancer Center (Other); Hospital Universitario Ramon y Cajal (Other); Hospital San Carlos, Madrid (Other); Centro Nacional de Investigaciones Oncologicas CARLOS III (Other)
Responsible Party: Sponsor-Investigator, Miguel Martín Jiménez, Professor of Medicine, Medical Oncology Service, Hospital General Universitario Gregorio Marañon
Organization: Hospital General Universitario Gregorio Marañon (Other)
Other Study IDs: GOMHGUGM022011
Record Dates: First submitted 2012-03-20; First posted 2012-03-22 (Estimated); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Breast Cancer; Breast Cancer Stage II-III
Keywords: Breast Cancer; Neoadjuvant therapy; Triple negative; predictor of response; predictor of resistance; Continuous Renal Replacement Therapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA and RNA from triple negative breast cancer patients
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Docetaxel Carboplatino: Doses of AUC 5-6 of carboplatin in combination with 75 mg/m2 of docetaxel are easily combined, being myelosuppression the most important toxicity. This combination has been studied in metastatic breast cancer as well as in the neoadjuvant setting. The combination of taxanes and platinum salts is increasingly used as neoadjuvant chemotherapy for TNBC. The docetaxel-carboplatin (TCb) regimen is an active and tolerable regimen in metastatic and locally advanced breast cancer, and the efficacy and toxicity characterization in the clinical setting are regaining interest in the era where the role of anthracyclines is controversial in the adjuvant setting. The avoidance of potentially serious long-term toxicities in specific breast cancer subtypes is a real challenge in an attempt to individualize therapies.
  Interventions: Drug: Docetaxel- Carboplatin

INTERVENTIONS:
Drug: Docetaxel- Carboplatin — Docetaxel 75mg/m2 day 1 and Carboplatin(AUC6)day 1, each 21 days for 6 cycles.

SUMMARY:
Neoadjuvant (preoperative) chemotherapy is an interesting research tool which allows investigators to test new drugs and/or new schedules with a validated surrogate endpoint, pCR. It also represents an ideal model to evaluate the relationships between treatments and tumor biomarkers. Recent publications have shown that new molecular classifications of breast cancer (intrinsic subtypes) have an important prognostic and predictive value. Using microarrays for gene expression profiling seems to be the best way to perform this classification; nevertheless such assays are not optimally available for common clinical practice. The IHC-based classification systems are still useful, as fresh tissue is not normally available in clinical practice, and has been shown to correlate well with intrinsic classification using gene expression microarrays. Recently the PAM50 gene set provided a risk of relapse score not only in ER-positive, node negative patients (similarly to the Oncotype Dx Recurrence Score) but also in the ER negative disease. Additionally, the PAM 50 assay was highly predictive of neoadjuvant response when considering all patients. This assay added significant prognostic and predictive value to pathologic staging, histologic grade, and standard clinical molecular markers while using an easy technique that can be performed in clinical practice because the qRT-PCR assay can be performed using FFEP tissue.

Triple Negative Breast Cancer (TNBC) is defined by a lack of expression of ER, PgR and HER-2. DNA microarray profiling studies have led to the classification of invasive breast carcinoma into five subtypes: luminal A and B, normal breast-like, HER2/neu overexpressing and basal-like subtypes, with clinical implications. Later on, a new subtype, the claudin-low, has been described. Although not synonymous, the majority of TNBCs carry the basal-like breast cancer (BLBC) molecular profile.

The triple negative subtype accounts for 11-20% of breast cancer in different studies, whereas in selected cohorts of patients with advanced breast cancer or African-American ethnicity, TNBC may be diagnosed among as many as 23-28%.

Patients with TN breast tumors treated with standard chemotherapy have a shorter DFS and OS than non-TNBC, this difference have been shown to be independent from tumor grade, nodal status and treatment in some studies. The peak risk of recurrence occurs within the first 3 years after initial treatment, with the majority of deaths occurring in the first five years.

Chemotherapy remains the only systemic treatment option available for TNBC patients. Several studies have shown that TNBC/BLBC is associated with an increased response rate to neoadjuvant chemotherapy when compared with luminal tumors. However, TNBC patients have a significantly decreased DFS and OS in comparison with luminal patients. The largest study exploring response and survival in early stage breast cancer treated with neoadjuvant chemotherapy was reported by Liedtke et al. Although an increase pCR rate was observed among the TNBC patients, they had a shorter lifespan than the non-TN ones. Patients experiencing pCR had an excellent OS regardless of hormone receptor expression, but patients with residual disease had a significantly shorter survival associated with TNBC compared with non-TN ones. This demonstrates that poor OS is derived from chemo-resistant patients (what unfortunately represent > 50% of them).

A relevant problem is the differential response to drugs of TN tumors. These tumors are usually treated with multidrug combinations including anthracyclines and taxanes, with pCR´s of 28-32%. Only recently, the results of a few small trials combining platinum salts and taxanes have been reported, with encouraging results (pCR of 44-77%). The taxane-platinum salt combinations have a biological background, since TN not associated BRCA1 mutations are sensitive to taxanes and resistant to anthracyclines and platinum salts are effective in TN tumors probably because a significant proportion of them have functional DNA repair deficiencies.

The primary objective of the study is to identify predictors of response to docetaxel-carboplatin in patients with triple negative primary tumors. Response is defined as lack of invasive tumor in breast plus axilla after neoadjuvant chemotherapy (PCR, pathological complete response).

DETAILED DESCRIPTION:
Neoadjuvant (preoperative) chemotherapy is an interesting research tool which allows investigators to test new drugs and/or new schedules with a validated surrogate endpoint, pCR. It also represents an ideal model to evaluate the relationships between treatments and tumor biomarkers. Recent publications have shown that new molecular classifications of breast cancer (intrinsic subtypes) have an important prognostic and predictive value. Using microarrays for gene expression profiling seems to be the best way to perform this classification; nevertheless such assays are not optimally available for common clinical practice. The IHC-based classification systems are still useful, as fresh tissue is not normally available in clinical practice, and has been shown to correlate well with intrinsic classification using gene expression microarrays. Recently the PAM50 gene set provided a risk of relapse score not only in ER-positive, node negative patients (similarly to the Oncotype Dx Recurrence Score) but also in the ER negative disease. Additionally, the PAM 50 assay was highly predictive of neoadjuvant response when considering all patients. This assay added significant prognostic and predictive value to pathologic staging, histologic grade, and standard clinical molecular markers while using an easy technique that can be performed in clinical practice because the qRT-PCR assay can be performed using FFEP tissue.

Triple Negative Breast Cancer (TNBC) is defined by a lack of expression of ER, PgR and HER-2. DNA microarray profiling studies have led to the classification of invasive breast carcinoma into five subtypes: luminal A and B, normal breast-like, HER2/neu overexpressing and basal-like subtypes, with clinical implications. Later on, a new subtype, the claudin-low, has been described. Although not synonymous, the majority of TNBCs carry the basal-like breast cancer (BLBC) molecular profile. The triple negative subtype accounts for 11-20% of breast cancer in different studies, whereas in selected cohorts of patients with advanced breast cancer or African-American ethnicity, TNBC may be diagnosed among as many as 23-28%. Patients with TN breast tumors treated with standard chemotherapy have a shorter DFS and OS than non-TNBC, this difference have been shown to be independent from tumor grade, nodal status and treatment in some studies. The peak risk of recurrence occurs within the first 3 years after initial treatment, with the majority of deaths occurring in the first five years.

Chemotherapy remains the only systemic treatment option available for TNBC patients. Several studies have shown that TNBC/BLBC is associated with an increased response rate to neoadjuvant chemotherapy when compared with luminal tumors. However, TNBC patients have a significantly decreased DFS and OS in comparison with luminal patients. The largest study exploring response and survival in early stage breast cancer treated with neoadjuvant chemotherapy was reported by Liedtke et al. Although an increase pCR rate was observed among the TNBC patients, they had a shorter lifespan than the non-TN ones. Patients experiencing pCR had an excellent OS regardless of hormone receptor expression, but patients with residual disease had a significantly shorter survival associated with TNBC compared with non-TN ones. This demonstrates that poor OS is derived from chemo-resistant patients (what unfortunately represent > 50% of them).

A relevant problem is the differential response to drugs of TN tumors. These tumors are usually treated with multidrug combinations including anthracyclines and taxanes, with pCR´s of 28-32%. Only recently, the results of a few small trials combining platinum salts and taxanes have been reported, with encouraging results (pCR of 44-77%). The taxane-platinum salt combinations have a biological background, since TN not associated BRCA1 mutations are sensitive to taxanes and resistant to anthracyclines and platinum salts are effective in TN tumors probably because a significant proportion of them have functional DNA repair deficiencies.

Role of anthracyclines and taxanes in TN breast cancer Efficacy results of anthracycline-based regimens in patients with TNBC remain controversial. The analysis from the MA5 study (which randomized patients between CMF and FEC), showed an increased 5-year DFS in favor of CMF (71% vs 51%) in the basal-like subtype group. The test for interaction between biologic phenotype and treatment arm almost reached significance (p=0,06) indicating that patients with TNBC may not derive a particular benefit from anthracyclines.

Several phase III studies comparing classical anthracycline schedules with anthracycline plus taxane treatment have performed retrospective analysis classifying patients between the different breast cancer subtypes. Results from those analysis showed that TNBC/BLBC patients treated with classic anthracycline regimens were having a very poor outcome (similar or in some of these studies even worse than the HER2 overexpressing patients before the trastuzumab era). In those studies the TNBC/BLBC populations were the ones benefiting the most from the taxane addition.

In addition to that, a single study by our group has compared single agent doxorubicin versus single agent docetaxel as neoadjuvant chemotherapy for locally advanced breast cancer. In this study, both drugs were similar in luminal and her2 subtypes, but docetaxel was significantly superior to doxorubicin in patients with basal-like tumors (good pathological response rate of 56% vs 0%, p=0.034). Besides, triple negative status was the only significant predictor of resistance to doxorubicin in multivariate analysis. Residual cancer burden after neoadjuvant chemotherapy in triple negative tumors was also significantly higher with doxorubicin than with docetaxel, thus indicating that this subtype is more resistant to doxorubicin than to docetaxel. This study firmly suggest that docetaxel should be the backbone of combination regimens for basal-like tumors and questions the role of doxorubicin in these tumors.

Role of platinum salts in TN breast cancer The role of platinum salts in TNBC is currently a matter of investigation. Basal-like breast cancers (BLBC) are highly aneuploid, associated with BRCA1 germline mutations, and have loss of TP53, RB1 and Chromosome 5q. None of these characteristics are observed in Claudin-low tumors suggesting a different etiology, and possibly, a different response to DNA damaging agents. Phase II studies have suggested that platinum salts have a significant activity en TNBC, particularly in BRCA-1 mutation carriers. Unfortunately, we cannot distinguish TNBC from Claudin-low with conventional IHC techniques.

Activity and side effects of the combination docetaxel-carboplatin in breast cancer The combination of carboplatin and docetaxel has been extensively studied mainly in ovarian and lung cancer. Doses of AUC 5-6 of carboplatin in combination with 75 mg/m2 of docetaxel are easily combined, being myelosuppression the most important toxicity. This combination has been studied in metastatic breast cancer as well as in the neoadjuvant setting.

Perez et al studied docetaxel (75 mg/m2 IV over 1 hour) followed by carboplatin (AUC 6 IV over 30 minutes) as first-line chemotherapy in 53 women with MBC. Patients received a median of 6 cycles. An overall response rate (ORR) of 60% (complete response [CR] 6%, partial response [PR] 54%) was noted. Grade 3/4 toxicities included anemia (11%), neutropenia (94%), thrombocytopenia (17%), febrile neutropenia (15%), leukopenia (15%), fatigue (21%), infection (11%), diarrhea (11%), hypersensitivity (8%), neurosensory (4%), and neuromotor (4%). A total of 26 patients received granulocyte colony-stimulating factor (G-CSF) and/or erythropoietin support. The authors concluded that although myelosuppression was noted, docetaxel and carboplatin were an active treatment regimen for first-line therapy in MBC and prophylactic hematopoietic growth factor support is recommended.

Docetaxel and carboplatin was evaluated in another phase II study in 40 patients with previously untreated MBC. Patients received docetaxel (75 mg/m2) and carboplatin (AUC 5) on day 1 every 3 weeks for up to 6 cycles. An ORR of 59% (CR 15.4%, PR 43.6%) was observed among the 39 patients evaluable for response. Grade 3/4 toxicities included neutropenia (n=28), febrile neutropenia (n=4), and thrombocytopenia (n=4). The authors concluded docetaxel and carboplatin were efficacious as first-line treatment for metastatic breast cancer, with an acceptable toxicity profile.

An additional phase II study with the same schedule was performed, as first-line chemotherapy in 32 patients (30 female, 2 male) with metastatic breast cancer. An ORR of 62.07% (8 CRs, 10 PRs) was reported; five patients (17.24%) had progressive disease. Grade 3 toxicities included neutropenia (24%), anemia (15.6%); nausea, vomiting, fluid retention, and peripheral neuropathy occurred in 15 patients. There were no reports of febrile neutropenia, nor were there any deaths. The authors concluded that the combination of docetaxel and carboplatin as first-line therapy in metastatic breast cancer patients was promising with well-tolerated toxicities. A fourth trial also with the same schedule determined the safety and efficacy of the combination in 25 women with MBC. An ORR of 56% (CR 24%, PR 32%) was reported. Grade 3/4 toxicities included neutropenia (24%), one case of febrile neutropenia that required hospitalization and two patients with diarrhea. Anemia noted in seven patients was deemed "mild" and there were no reported toxic deaths. The authors concluded combination docetaxel and carboplatin was safe and active as first-line therapy in patients with MBC.

With regards to its use in the neoadjuvant treatment, this combination was studied in 57 patients with stage II/III breast cancer (10). Docetaxel (75 mg/m2) and carboplatin (AUC 6) were given on day 1 with pegfilgrastim (6 mg subcutaneously) on day 2. This regimen was repeated in a dose-dense manner every 2 weeks for 4 cycles. Fifty-one patients (89%) had breast-conserving surgery within 6 weeks. Among all 57 patients, a pathological complete response (pCR) of 16% was reported. Four out of 9 patients with triple negative tumors had pCR (44%). Thrombocytopenia was the only grade 4 toxicity reported. Grade 3 toxicities in addition to thrombocytopenia consisted of anemia, fatigue, diarrhea, nausea, and hypokalemia. The authors concluded the combination of docetaxel, carboplatin, and pegfilgrastim was feasible and tolerable in all patients.

In a phase II trial, Karmarkar et al investigated a neoadjuvant regimen of four cycles of docetaxel (90 mg/m2) and carboplatin (AUC 6) on day 1 with filgrastim every 3 weeks in 22 patients with locally advanced breast cancer. After four cycles, patients underwent surgery. A total of 16 patients were evaluable for efficacy and toxicity. There were five complete responses and 11 partial responses reported. Grade 3/4 toxicities included myelosuppression with infection (n=1), myalgia (n=2), diarrhea (n=1), fatigue/asthenia (n=5), and nausea (n=4). The authors concluded that this neoadjuvant combination of docetaxel and carboplatin was active and well tolerated; they also noted that the addition of filgrastim allowed a dose intense regimen to be delivered.

A recently published phase II performed by Chang et al studied the same regimen but with a lower docetaxel dose (75 mg/m2) and without G-CSF support. Seventy-three patients were treated for 4 cycles (11 of them were TNBC). Patients HER2 positive were additionally randomized to chemotherapy alone or in combination with trastuzumab weekly. Seventy-one patients underwent surgery from which 19 (26.8%) had pCR (absence of invasive breast cancer in the breast), 6 of them within the TNBC subgroup. Grade 3/4 toxicities other than hematological, such as neutropenia (43%), and febrile neutropenia (4%) were rare. Grade 3 docetaxel hypersensitivity was noted in 4% of patients and all other grade 3/4 adverse events occurred in less than 2% of them.

All shown data, together with the potential anthracycline cardiotoxicity and risk of anthracycline-induced leukemias in patients with a high probability of being cured, challenge the role of anthracyclines in the treatment of early stage TNBC patients. The combination of taxanes and platinum salts is, therefore, increasingly used as neoadjuvant chemotherapy for triple negative breast cancer. The docetaxel-carboplatin (TCb) regimen is an active and tolerable regimen in metastatic and locally advanced breast cancer, and the efficacy and toxicity characterization in the clinical setting are regaining interest in the era where the role of anthracyclines is controversial in the adjuvant setting. The avoidance of potentially serious long-term toxicities in specific breast cancer subtypes is a real challenge in an attempt to individualize therapies.

In the daily practice, however, we have problems identifying basal-like tumors, since not all triple negative tumors belongs to this subtype. We need, therefore, predictive markers of response to neoadjuvant chemotherapy in general and the docetaxel-carboplatin regimen in particular.

STUDY OBJECTIVES:

Primary Objective The primary objective of the study is to identify predictors of response to docetaxel-carboplatin in patients with triple negative primary tumors. Response is defined as lack of invasive tumor in breast plus axilla after neoadjuvant chemotherapy (PCR, pathological complete response).

Secondary Objective(s)

Secondary objectives are the following:

* To identify predictors of good pathological response according to Symmans criteria (i.e. Symmans class 0+1).
* To identify predictors of chemoresistance (class III od Symmans)
* To assess the clinical response rate by standard methods (MRI, clinical examination, mammogram) in patients treated with this regimen.
* To evaluate breast conserving surgery rate in patients treated with this regimen.
* To evaluate the pCR rate in patients with known BRCA mutations.

STUDY DESIGN:

Patients with triple negative tumors according to a core biopsy scheduled to be treated with docetaxel plus carboplatin (i.e., no contraindications for the regimen) will be candidate for the study. After detailed information of study purposes, they will be asked to sign an informed consent Triple negative status is defined as ER <1% stained cells, PR <1% stained cells and HER2 negative (IHC of 0-1+ or or 2-3+ with FISH/CISH negative testing).

Patients will have 6 cycles of docetaxel (75 mg/m2 IV day 1) plus carboplatin (AUC 6, IV day 1) every 3 weeks (TCb regimen). Patients with objective response or stable disease will undergo surgery after the sixth cycle.

While on treatment, patients will be assessed as clinically indicated to discard progression with breast MRI. A biopsy will be performed to confirm progression and the patient will be removed from the study and treated according to investigator's criteria, usually with anthracycline-containing regimens (i.e. FE90C, 5FU 600 mg/m2 IV, epirubicin 90 mg/m2 IV, cyclophosphamide 600 mg/m2 IV, day 1 every 3 weeks).

Patients who achieve a pathological complete response at surgery will not receive additional chemotherapy (radiation therapy will be administered as indicated by local criteria, i.e., breast preserving surgery, large tumors >5 cm, axillary involvement). Those patients who do not achieve a pathological complete response at surgery will receive 3 additional cycles of FE90C chemotherapy after the surgical procedure.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent form signed by the patient to accept study enrollment.
* Female with pathologically confirmed diagnosis of primary invasive operable breast cancer, stage IIa-IIIc (6th edition of the AJCC Cancer Staging Manual), with tumors ≥ 2cm.

Triple negative phenotype patients (RE and PR of less than 1% of stained cells by IHQ, IHC for HER2 of 0-1+ or ISH negative if 2/3+), according to local laboratory.

* Age 18-75 years.
* Adequate performance status (ECOG <2).
* Adequate renal and liver function and bone marrow reserve.

Exclusion Criteria:

* Clinical or radiologic evidence of Metastatic disease.
* Prior or concurrent anti-cancer therapy for current disease (hormone therapy, chemotherapy, radiotherapy, immunotherapy).
* Prior therapy with taxanes, anthracyclines or carboplatin for any malignancy.
* Contraindication for study drugs (docetaxel or carboplatin).
* Serious concomitant systemic disorder that in the opinion of the investigator would compromise the patient's ability to complete the study, or have any other disease that could be worsened by chemotherapy or other potential support therapies.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female patients with triple negative primary tumors
Sampling Method: Non-Probability Sample
Enrollment: 415 (Estimated)
Dates: Start 2012-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
predictors of response to docetaxel-carboplatin in patients with triple negative primary tumors | 6 months
  The primary objective of the study is to identify predictors of response to docetaxel-carboplatin in patients with triple negative primary tumors. Response is defined as lack of invasive tumor in breast plus axilla after neoadjuvant chemotherapy (PCR, pathological complete response).

SECONDARY OUTCOMES:
predictors of good pathological response and chemoresistance | 3 months
  * To identify predictors of good pathological response according to Symmans criteria (i.e. Symmans class 0+1)
  * To identify predictors of chemoresistance (class III od Symmans)
  * To assess the clinical response rate by standard methods (MRI, clinical examination, mammogram) in patients treated with this regimen.
  * To evaluate breast conserving surgery rate in patients treated with this regimen.
  * To evaluate the pCR rate in patients with known BRCA mutations.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Gregorio Marañon, Madrid, Spain

REFERENCES:
- [Background] Echavarria I, Lopez-Tarruella S, Picornell A, Garcia-Saenz JA, Jerez Y, Hoadley K, Gomez HL, Moreno F, Monte-Millan MD, Marquez-Rodas I, Alvarez E, Ramos-Medina R, Gayarre J, Massarrah T, Ocana I, Cebollero M, Fuentes H, Barnadas A, Ballesteros AI, Bohn U, Perou CM, Martin M. Pathological Response in a Triple-Negative Breast Cancer Cohort Treated with Neoadjuvant Carboplatin and Docetaxel According to Lehmann's Refined Classification. Clin Cancer Res. 2018 Apr 15;24(8):1845-1852. doi: 10.1158/1078-0432.CCR-17-1912. Epub 2018 Jan 29. PMID 29378733
- [Background] Sharma P, Lopez-Tarruella S, Garcia-Saenz JA, Khan QJ, Gomez HL, Prat A, Moreno F, Jerez-Gilarranz Y, Barnadas A, Picornell AC, Monte-Millan MD, Gonzalez-Rivera M, Massarrah T, Pelaez-Lorenzo B, Palomero MI, Gonzalez Del Val R, Cortes J, Fuentes-Rivera H, Morales DB, Marquez-Rodas I, Perou CM, Lehn C, Wang YY, Klemp JR, Mammen JV, Wagner JL, Amin AL, O'Dea AP, Heldstab J, Jensen RA, Kimler BF, Godwin AK, Martin M. Pathological Response and Survival in Triple-Negative Breast Cancer Following Neoadjuvant Carboplatin plus Docetaxel. Clin Cancer Res. 2018 Dec 1;24(23):5820-5829. doi: 10.1158/1078-0432.CCR-18-0585. Epub 2018 Jul 30. PMID 30061361
- [Background] Picornell AC, Echavarria I, Alvarez E, Lopez-Tarruella S, Jerez Y, Hoadley K, Parker JS, Del Monte-Millan M, Ramos-Medina R, Gayarre J, Ocana I, Cebollero M, Massarrah T, Moreno F, Garcia Saenz JA, Gomez Moreno H, Ballesteros A, Ruiz Borrego M, Perou CM, Martin M. Breast cancer PAM50 signature: correlation and concordance between RNA-Seq and digital multiplexed gene expression technologies in a triple negative breast cancer series. BMC Genomics. 2019 Jun 3;20(1):452. doi: 10.1186/s12864-019-5849-0. PMID 31159741
- [Background] Yau C, Osdoit M, van der Noordaa M, Shad S, Wei J, de Croze D, Hamy AS, Lae M, Reyal F, Sonke GS, Steenbruggen TG, van Seijen M, Wesseling J, Martin M, Del Monte-Millan M, Lopez-Tarruella S; I-SPY 2 Trial Consortium; Boughey JC, Goetz MP, Hoskin T, Gould R, Valero V, Edge SB, Abraham JE, Bartlett JMS, Caldas C, Dunn J, Earl H, Hayward L, Hiller L, Provenzano E, Sammut SJ, Thomas JS, Cameron D, Graham A, Hall P, Mackintosh L, Fan F, Godwin AK, Schwensen K, Sharma P, DeMichele AM, Cole K, Pusztai L, Kim MO, van 't Veer LJ, Esserman LJ, Symmans WF. Residual cancer burden after neoadjuvant chemotherapy and long-term survival outcomes in breast cancer: a multicentre pooled analysis of 5161 patients. Lancet Oncol. 2022 Jan;23(1):149-160. doi: 10.1016/S1470-2045(21)00589-1. Epub 2021 Dec 11. PMID 34902335
- See also: Related Info — http://doi.org/10.1186/s12864-019-5849-0
- See also: Related Info — http://doi.org/10.1016/S1470-2045(21)00589-1